CLINICAL TRIAL: NCT06918106
Title: Screening and Brief-Intervention of Post-war Alcohol Consumption in Public Hospital Outpatients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aksum University (Other)
Responsible Party: Principal Investigator, Abraha Gosh, PhD (Assistant Professor), Aksum University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AKU/CHS-CSH/MS/06/17
Record Dates: First submitted 2025-01-28; First posted 2025-04-09 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Effectiveness of Screening and Brief-Intervention; Unhealthy Alcohol Use
Keywords: Post-war alcohol use; Screening and Brief-intervention; Harmful alcohol use; Hazardous alcohol use

STUDY DESIGN:
Masking Description: Masking Description
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Control Group (Other): Participants in this group will not receive the intervention (Simple advice, Brief-counseling and broacher) except the screening for alcohol consumptions that will take at baseline (T1) and at 6 months (T2) and 12 months (T3) of follow-ups.
  Interventions: Behavioral: Simple advice, Brief-counseling and brochure

INTERVENTIONS:
Behavioral: Simple advice, Brief-counseling and brochure — Participants assigned to the intervention group will receive "simple advice" plus "brief counseling" and "health broacher" and then they will be screened for alcohol consumption at 6 months and 12 months of follow-ups.

SUMMARY:
Background:

High prevalence of alcohol-consumption among conflict-affected population has been reported in some low-and-middle income countries. However, studies that assess the effectiveness of screening and brief-intervention (SBI) in the reduction of unhealthy alcohol consumptions among conflict-affected hospital outpatients in Tigray are insufficient.

Objective:

This study aims to test the effectiveness of Screening and Brief-Intervention (SBI) in the reduction of unhealthy alcohol consumptions among conflict-affected hospital outpatients in Tigray.

Method:

About 1260 outpatients will be screened for alcohol consumption using Alcohol Use Disorder Identification Test (AUDIT). Those who will have "8-19" scores in the AUDIT will be allocated to "Intervention" and "Control" groups using block randomization and they will be followed at 6 and 12 months of follow - up. The Intervention group will receive simple advice, brief-counseling and 6-and 12-months follow-up screening of alcohol consumptions. However, outpatients in control group will only receive 6- and 12-months follow-up screening of alcohol consumptions. Data will be entered to and will be analyzed using SPSS V 26. Means, standard deviations and percentages will be used for descriptive statistics. Bivariate and multivariate logistic regression, at 95% of confidence interval and p-value of <0.05, will be used to identify correlates of alcohol consumption. Independent sample t-test and Mann-Whitney U test will be used to compare AUDIT mean scores of normally and none-normally distributed continuous variables between intervention and control groups respectively.

DETAILED DESCRIPTION:
Rationale:

Evidence on the effectiveness of screening and brief-intervention of unhealthy alcohol consumption in conflict-affected population in countries like Ethiopia are insufficient. This can affect the development and implementation of effective alcohol policies and interventions unless more studies strive to fill such gaps.

By screening post-war alcohol consumption and examining the efficacy of brief-interventions, this research will address the gap on the effectiveness of Screening and Brief-Intervention on reduction of hazardous/harmful alcohol consumption among public hospital outpatients. Findings can lead policymakers and health professionals to develop initiatives that promote abstinence or low risk drinking behavior to improve alcohol related health outcomes among hospital outpatients. Findings of this study can assist the development of evidence-based policy and management programs to reduce risky alcohol consumptions among public hospital outpatients.

Therefore, post-war alcohol consumption in Tigray public hospital outpatients needs to be rigorously studied to formulate an appropriate and effective intervention mechanism to prevent and reduce risky alcohol consumption among outpatients.

General Objectives:

To screen post-war alcohol consumptions and test the effectiveness of Brief-Intervention in reducing risky alcohol consumption among Public Hospital outpatients in Tigray from 2024 to 2026.

Specific Objectives:

To assess rate of post-war alcohol consumption among public hospital outpatients in Tigray from 2024 to 2026.

To determine associated factors of post-war alcohol consumptions among public hospital outpatients in Tigray from 2024 to 2026.

To test the effectiveness of screening and Brief-Intervention of alcohol consumption among public hospital outpatients in Tigray.

Methodology:

The researchers want to study the effectiveness of screening and brief-intervention of post-war alcohol consumption among public hospital outpatients in Tigray. The study will have a continuous outcome (AUDIT score) and equal sample size in both intervention and control groups. Therefore, the researchers prefer to use the simplest established formula to calculate the sample size in each group as follows.

Assuming the mean difference in AUDIT score between intervention and control groups that this study will bring is 4.4, Standard Deviation is 10, alpha (α) is 0.05 at 95% confidence interval, beta (β) is 0.20 then the sample size in each group is calculated to be n=81 with a total required sample of 162. However, since evidence are reporting that there were 28% and 33% of loss of follow-up at 6 and 12 months respectively, the required sample size in each group will be inflated to 131 with a total required sample size of 262. All female and male outpatients aged 18 years and above with no serious medical or mental illnesses with an AUDIT score of 8-19 will be included in the intervention. While outpatients less than 18 years, those with serious illnesses and have an AUDIT score of less than 7 or ≥ 20 will be excluded from the intervention.

Intervention group will receive a single session of simple advice, brief-counseling and broacher with 6-and 12-months follow-up screening. Whereas outpatients in control group will only receive the 6- and 12-months follow-up screening to see their level of alcohol consumption.

Data management and analysis Data will be collected via face-to-face interview by trained data collectors. Collected data will be handled in a secured place and in a confidential way. The data will be coded, entered and analyzed to SPSS Vs 26. Means, standard deviations and percentage will be used for the descriptive statistics. Independent sample t-test or Mann-Whitney U test will be used to compare the mean of normally distributed or none-normally distributed AUDIT scores between intervention and control groups respectively. Repeated measure ANOVA will be used to test the effectiveness of Screening and Brief-Intervention of post-war alcohol consumption. However, non-parametric alternatives like Friedman test will be also used if assumptions for parametric statistics are failed.

ELIGIBILITY:
Inclusion Criteria:

* All gender (Female & Male patients)
* Outpatients aged 18 years and above
* Outpatients with no serious medical or mental illnesses
* Outpatients who will be identified to have AUDIT score of 8-19

Exclusion Criteria:

* Age less than 18 years
* Outpatients with serious medical or mental illnesses
* Outpatients with AUDIT score of less than 7 and above 20

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 262 (Estimated)
Dates: Start 2025-04-03 (Actual); Primary Completion 2026-04-03 (Estimated); Study Completion 2026-04-03 (Estimated)

PRIMARY OUTCOMES:
Screening and brief-intervention of post-war Alcohol Use among hospital outpatpatients | Time frame schedule: 12 months
  Time one (T1) screening using Alcohol use disorders identification test (AUDIT) will identify
  1. study subjects with 0-7 AUDIT score which is equivalent to "Low Risk Drink" and will be excluded from the intervention.
  2. study subjects with 8-19 AUDIT score which is equivalent to "Hazardous/ Harmful Drink" and will enter to the brief-intervention.
  3. study subjects with 20 or more AUDIT score is equivalent to "Posible Alcohol dependency" and will be excluded from the study but referred for diagnostic evaluation and treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Suhul General Hospital: is a general hospital located in Shire Endasilassie town, Northwest Tigray. Suhul Hospital provides a wide range of medical services for more than 18,000 people every month and has a psychiatry outpatient department, Shirē, Tigray, Ethiopia

IPD SHARING:
Plan to Share IPD: No